CLINICAL TRIAL: NCT01952314
Title: Medical Expulsive Therapy for Ureter Stone Using Naftopidil: Multicenter, Randomized, Double-blind, Placebo Controlled Study
Brief Title: Medical Expulsive Therapy for Ureter Stone Using Naftopidil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chang Wook Jeong, M.D, Ph.D., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUBH-URO-2012-03; SNUBH-URO-2012-03-MET (Other: SNU Bundang Hospital IRB)
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Ureter Stones
MeSH Terms: interventions — naftopidil; Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control groups with only analgesics (Placebo Comparator): Control groups will receive only analgesics.
  Interventions: Drug: Placebo for Naftopidil; Drug: Standard treatment
- Naftopidil (Active Comparator): This interventional group will receive analgesics and naftopidil 75mg po qd.
  Interventions: Drug: Naftopidil 75mg; Drug: Standard treatment

INTERVENTIONS:
Drug: Naftopidil 75mg — naftopidil 75mg 1T qd hs
  Other Names: Flivas(TM) in South Korea
  Arms: Naftopidil
Drug: Placebo for Naftopidil — Placebo 1T qd hs
  Arms: Control groups with only analgesics
Drug: Standard treatment — Aceclofenac 100mg or tramadol37.5mg/acetaminophen 325mg on demand
  Other Names: Pain control

SUMMARY:
This study is to investigate whether naftopidil is effective or not for the spontaneous passage of ureteral stones with sizes of 3 to 10 mm.

DETAILED DESCRIPTION:
1. Enrollment

   1. patients with ureteral stones of sizes from 3 to 10 mm
   2. patients aged more than 18 years
2. Randomization

   1. naftopidil 75 mg qd for 14 days or placebo
   2. Standard treatment with pain-killers were also applied.(aceclofenac)
3. Follow-up for 28 days

   1. We confirm the stone free status by CT or X-ray films at 14th and 28th days.
   2. Rates of active treatment will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* >= 20 years
* single 3 to 10 mm ureter stone (longest diameter)

Exclusion Criteria:

* Presence of multiple ureter stones
* Renal insufficiency (serum Cr > 1.4 mg/dL)
* Febrile urinary tract infections(fever > 38°C, evidence of urinary infection)
* pregnancy or breast feeding
* solitary kidney
* hypersensitivity to naftopidil
* current use of any alpha-blocker, calcium-channel blocker, corticosteroid (within 4 weeks)
* moderate or severe cardiovascular or cerebrovascular disease
* hepatic dysfunction (>2 x normal upper limit)
* significant active medical illness which in the opinion of the investigator would preclude protocol treatment
* Genetic disorder such as Galactose intolerance, Lapp Lactase deficiency, Glucose-Galactose malabsorption

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Stone-free rate at 14th day of study | 14th day
  Rate of stone-free as confirmed by non-contrast CT, intravenous urography or simple x-ray (only for radio-opaque stone)

SECONDARY OUTCOMES:
Stone-free rate at 28th day of study | 28th day
Duration to stone passage within 28days of study | for 28 days
amount of analgesics used for 28 days of study | for 28 days
Rate of active treatment | for 28 days
  Active treatments include shock-wave lithotripsy, ureteroscopic ureterolithotomy, ureteral stenting or other surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chang Wook Jeong, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - Donguk University Ilsan Hospital, Goyang, Kyunggi
  - Seoul National University Bundang Hospital, Seongnam, Kyunggi
  - Kangwon National University Hospital, Chuncheon
  - Seoul National University Hospital, Seoul
  - National Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul